CLINICAL TRIAL: NCT01182558
Title: The Effect of Prior Muscle Activation on the Compound Muscle Action Potential (CMAP)- Implications for Routine Nerve Conduction Studies (NCS) and Serial NCS
Brief Title: The Effect of Prior Muscle Activation on the Compound Muscle Action Potential (CMAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Gordon Peterson, Professor of Neurology, Loma Linda University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 5100161
Record Dates: First submitted 2010-08-12; First posted 2010-08-17 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Focus: Effect of Muscle Activation on CMAP in Normal Humans
Keywords: Muscle; Activation; Effect; Compound muscle action potential
MeSH Terms: interventions — Neuromuscular Blockade

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Activation of Hypothenar Eminence (Other): Each subject will perform maximum, voluntary, isometric muscle activation (of the target muscle) for each of various lengths of time ("single brief muscle twitch," 2 seconds, 5 seconds, 10 seconds, and 20 seconds [two epochs of 10 seconds of muscle activation with 1-2 seconds of rest between the two epochs]).
  Interventions: Other: Hypothenar muscle activation--maximum, voluntary, isometric
- Activation of Thenar Eminence (Other): Each subject will perform maximum, voluntary, isometric muscle activation (of the target muscle) for each of various lengths of time ("single brief muscle twitch," 2 seconds, 5 seconds, 10 seconds, and 20 seconds [two epochs of 10 seconds of muscle activation with 1-2 seconds of rest between the two epochs]).
  Interventions: Other: Thenar muscle activation--maximum, voluntary, isometric
- Activation of Extensor Digitorum Brevis (Other): Each subject will perform maximum, voluntary, isometric muscle activation (of the target muscle) for each of various lengths of time ("single brief muscle twitch," 2 seconds, 5 seconds, 10 seconds, and 20 seconds [two epochs of 10 seconds of muscle activation with 1-2 seconds of rest between the two epochs]).
  Interventions: Other: EDB muscle activation--maximum, voluntary, isometric
- Maintain Relaxation of the Opposite Side (Placebo Comparator): While the muscle of the right side is activated periodically and the compound muscle action potential is tested frequently, the muscle on the left side is maintained at rest and the compound muscle action potential is tested infrequently.
  Interventions: Other: Relaxation of muscle

INTERVENTIONS:
Other: Hypothenar muscle activation--maximum, voluntary, isometric — Each subject will perform maximum, voluntary, isometric muscle activation (of the target muscle) for each of various durations ("single brief muscle twitch," 2 seconds, 5 seconds, 10 seconds, and 20 seconds [two epochs of 10 seconds of muscle activation with 1-2 seconds of rest between the two epochs]).
  Arms: Activation of Hypothenar Eminence
Other: Thenar muscle activation--maximum, voluntary, isometric — Each subject will perform maximum, voluntary, isometric muscle activation (of the target muscle) for each of various durations ("single brief muscle twitch," 2 seconds, 5 seconds, 10 seconds, and 20 seconds [two epochs of 10 seconds of muscle activation with 1-2 seconds of rest between the two epochs]).
  Arms: Activation of Thenar Eminence
Other: EDB muscle activation--maximum, voluntary, isometric — Each subject will perform maximum, voluntary, isometric muscle activation (of the target muscle) for each of various durations ("single brief muscle twitch," 2 seconds, 5 seconds, 10 seconds, and 20 seconds [two epochs of 10 seconds of muscle activation with 1-2 seconds of rest between the two epochs]).
  Arms: Activation of Extensor Digitorum Brevis
Other: Relaxation of muscle — The muscle on the opposite side will be maintained at rest.
  Arms: Maintain Relaxation of the Opposite Side

SUMMARY:
The purpose of this investigator-initiated study is to determine the effect of prior muscle activation on the response obtained by nerve conduction studies (the compound muscle action potential [CMAP]) looking at the amplitude, area, and duration of the CMAP and evaluating the length of time the CMAP is larger than at baseline. On the opposite side, the corresponding CMAP will be tested periodically, but there will be no muscle activation on that side.

Null Hypothesis: While controlling all possible technical and other known physiological variables, prior activation of a muscle has no effect on the amplitude and area of the compound muscle action potential (CMAP); and the CMAP does not change over time in the relaxed muscle (on the opposite side).

The investigators suspect that there is an effect of prior activation of the muscle on the subsequent CMAP recorded from that muscle.

DETAILED DESCRIPTION:
Nerve conduction studies (NCS) will be performed with supramaximal nerve stimulation, surface stimulation, surface recording, and with best possible technique controlling as many variables as possible including the location of the recording electrodes and with a warm muscle and nerve (measuring temperature at the skin) in each of 3 "arms" of the study:

* ulnar nerve stimulation at the wrist recording from the hypothenar eminence,
* median nerve stimulation at the wrist recording from the thenar eminence, and
* peroneal nerve stimulation at the ankle recording from the extensor digitorum brevis muscle.

NCS will be performed in a rested muscle (rested for 15 minutes or longer) and then multiple times for up to 40 minutes after maximum isometric contraction (activation) of the tested muscle for a defined length of time. The defined lengths of muscle activation include:

* "a brief twitch" (activation for a fraction of a second),
* 2 seconds,
* 5 seconds,
* 10 seconds, and
* 20 seconds (two epochs of 10 seconds of activation with 1-2 seconds of rest between the two epochs).

The CMAP will be recorded multiple times from the muscle which was activated (pre-activation; as well as post-activation at multiple times after muscle activation: immediately, 5 sec, 10 sec, 15 sec, 20 sec, 30 sec, 60 sec, 90 sec, 2 minutes, and every minute up to as long as 40 minutes). Similar recordings will be made after each of the 5 durations of muscle activation ("a brief twitch," 2 seconds, 5 seconds, 10 seconds, and 20 seconds) of each of the three muscles (hypothenar, thenar, and EDB). CMAP amplitude (baseline to negative peak), area (under the negative curve), and duration (of the negative CMAP) will each be measured at each timepoint; and skin temperature in the region of the "active" recording electrode will be measured. Each data type will be compared over time in a series, identified as muscle from which recorded, duration of muscle activation performed prior to the recording, and time after the end of muscle activation.

On a few occasions during the testing of the CMAP on the side on which the muscle is activated, there will be recording of the CMAP from the corresponding muscle on the opposite side, but that second side will be relaxed the entire time of testing (for 4-5 hours).

If the CMAP changes more than a small amount on either side, F waves may be tested while the muscle is at rest.

Each subject will participate in each of the 3 "arms." Testing for the five series of recordings from each muscle is anticipated to take 4-5 hours, i.e., after screening, 12-15 hours total for testing the 3 muscles in each subject.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy volunteers
* Age 18-49

Exclusion Criteria:

* Localized or generalized neuromuscular disorder
* History of neuropathy
* History of diabetes
* History of prior injuries or surgeries of the back, neck, or limbs to be tested which in the opinion of the investigator might have the potential to influence the compound muscle action potential
* Medications other than eyedrops or non-steroidal anti-inflammatory agents (as needed) or contraceptive agents or non-steroidal topical agents
* Abnormalities by screening nerve conduction studies
* Anomalous innervation of the tested extensor digitorum brevis via screening nerve conduction studies
* Use of caffeine or nicotine within 8 hours of testing

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Ulnar-Hypothenar CMAP Amplitude | Immediate, 5 sec, 10 sec, 15 sec, 20 sec, 30 sec, 60 sec, 90 sec, 2 minutes, and each minute up to 40 minutes (or return to pre-activation value)
  Amplitude (baseline to negative peak) of the compound muscle action potential (CMAP) recorded from the hypothenar eminence after stimulation of the ulnar nerve at the wrist
Ulnar-Hypothenar CMAP Area | Immediate, 5 sec, 10 sec, 15 sec, 20 sec, 30 sec, 60 sec, 90 sec, 2 minutes, and each minute up to 40 minutes (or return to pre-activation value)
  Area (under the negative curve) of the compound muscle action potential (CMAP) recorded from the hypothenar eminence after stimulation of the ulnar nerve at the wrist
Median-Thenar CMAP Amplitude | Immediate, 5 sec, 10 sec, 15 sec, 20 sec, 30 sec, 60 sec, 90 sec, 2 minutes, and each minute up to 40 minutes (or return to pre-activation value)
  Amplitude (baseline to negative peak) of the compound muscle action potential (CMAP) recorded from the thenar eminence after stimulation of the median nerve at the wrist
Median-Thenar CMAP Area | Immediate, 5 sec, 10 sec, 15 sec, 20 sec, 30 sec, 60 sec, 90 sec, 2 minutes, and each minute up to 40 minutes (or return to pre-activation value)
  Area (under the negative curve) of the compound muscle action potential (CMAP) recorded from the thenar eminence after stimulation of the median nerve at the wrist
Peroneal-EDB CMAP Amplitude | Immediate, 5 sec, 10 sec, 15 sec, 20 sec, 30 sec, 60 sec, 90 sec, 2 minutes, and each minute up to 40 minutes (or return to pre-activation value)
  Amplitude (baseline to negative peak) of the compound muscle action potential (CMAP) recorded from the extensor digitorum brevis muscle (EDB) after stimulation of the peroneal nerve at the ankle
Peroneal-EDB CMAP Area | Immediate, 5 sec, 10 sec, 15 sec, 20 sec, 30 sec, 60 sec, 90 sec, 2 minutes, and each minute up to 40 minutes (or return to pre-activation value)
  Area (under the negative curve) of the compound muscle action potential (CMAP) recorded from the extensor digitorum brevis muscle (EDB) after stimulation of the peroneal nerve at the ankle

SECONDARY OUTCOMES:
Ulnar-Hypothenar CMAP Duration | Immediate, 5 sec, 10 sec, 15 sec, 20 sec, 30 sec, 60 sec, 90 sec, 2 minutes, and each minute up to 40 minutes (or return to pre-activation value)
  Duration (of the negative curve) of the compound muscle action potential (CMAP) recorded from the hypothenar eminence after stimulation of the ulnar nerve at the wrist
Median-Thenar CMAP Duration | Immediate, 5 sec, 10 sec, 15 sec, 20 sec, 30 sec, 60 sec, 90 sec, 2 minutes, and each minute up to 40 minutes (or return to pre-activation value)
  Duration (of the negative curve) of the compound muscle action potential (CMAP) recorded from the thenar eminence after stimulation of the median nerve at the wrist
Peroneal-EDB CMAP Duration | Immediate, 5 sec, 10 sec, 15 sec, 20 sec, 30 sec, 60 sec, 90 sec, 2 minutes, and each minute up to 40 minutes (or return to pre-activation value)
  Duration (of the negative curve) of the compound muscle action potential (CMAP) recorded from the extensor digitorum brevis muscle (EDB) after stimulation of the peroneal nerve at the ankle
Size of the CMAP from the Contralateral Limb Muscle While at Rest | Record periodically (every 1-15 minutes)
  The amplitude, area, and duration of the compound muscle action potential (CMAP) recorded from the contralateral muscle (Ulnar-Hypothenar, Median-Thenar, or Peroneal-EDB) will be determined as this contralateral muscle stays at rest.
F Wave Size and Persistence | Periodically
  F waves may be determined and the size and persistence of the F wave may be determined at baseline and if the amplitude of the direct response recorded from the muscle (on either the side of muscle activation or the side continuing at rest) with nerve stimulation changes by more than a small amount.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon W. Peterson, MD, Principal Investigator — Neurology, Faculty Physicians and Surgeons of Loma Linda University School of Medicine
Locations (1):
- Neurology - Faculty Physicians and Surgeons of Loma Linda University School of Medicine, Loma Linda, California, United States

REFERENCES:
- [Background] Peterson GW, Tsao BE, Nist LD, Estevez D, Brandstater ME. Prior muscle activation affects the compound muscle action potential. Muscle Nerve. 2019 Jul;60(1):25-31. doi: 10.1002/mus.26463. Epub 2019 Mar 25. PMID 30847939